CLINICAL TRIAL: NCT03492554
Title: Electrocardiogram Clinical Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apple Inc. (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 099-11774
Record Dates: First submitted 2018-02-27; First posted 2018-04-10 (Actual); Results first posted 2019-07-24 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Atrial fibrillation (AF) (Other): Patient with a known history of AF who are in AF at the time of study screening.
  Interventions: Other: 1-Lead ECG; Device: 12-Lead ECG
- Normal Sinus Rhythm (SR) (Other): Patient with no known diagnosis of AF or other arrhythmia
  Interventions: Other: 1-Lead ECG; Device: 12-Lead ECG

INTERVENTIONS:
Other: 1-Lead ECG — All participants will record three single-lead ECGs
Device: 12-Lead ECG — All participants will simultaneously record three 12-lead ECGs

SUMMARY:
The purpose of the study is to confirm the software's ability to create a Lead-1 electrocardiogram (ECG) that is clinically equivalent to a reference device. Also, to confirm a rhythm classification algorithm and its ability to detect and classify heart rhythms into two categories (Sinus Rhythm or Atrial Fibrillation) using a single Lead ECG.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are 22 years of age and older
* Able to read, understand, and provide written informed consent
* Willing and able to participate in the study procedures as described in the consent
* Have a wrist circumference that fits within the band
* Able to communicate effectively with and follow instructions from the study staff
* For subjects enrolled into the AF population, subjects must have a known diagnosis of AF and be in AF at the time of screening

Exclusion Criteria:

* Physical disability that precludes safe and adequate testing
* Mental impairment resulting in limited ability to cooperate
* Subjects with a pacemaker or implantable cardioverter-defibrillator (ICD)
* Acute myocardial infarction (MI) within 90 days of screening or other cardiovascular disease that, in the opinion of the Investigator, increases the risk to the subject or renders data uninterpretable
* Acute pulmonary embolism, pulmonary infarction, or deep vein thrombosis within 90 days of screening
* Stroke or transient ischemic attack within 90 days of screening
* Subjects taking rhythm control drugs
* Symptomatic (or active) allergic skin reactions such as eczema, rosacea, impetigo, dermatomyositis or allergic contact dermatitis on both wrists or over electrode attachment sites
* Known sensitivity to medical adhesives, isopropyl alcohol, watch bands, or electrocardiogram (ECG) electrodes including known allergy or sensitivity to fluoroelastomer bands primarily used in wrist worn fitness devices
* A history of abnormal life-threatening rhythms as determined by the investigator
* Significant tremor that prevents subject from being able to hold still
* Pregnant women: Women who are pregnant at the time of study participation
* For subjects enrolled into the sinus rhythm population, they must not have any diagnosis of AF

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-05-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - QPS, Miami, Florida
  - BioClinicia- Orlando, Orlando, Florida
  - BioClinica- The Villages, The Villages, Florida
  - IQVIA, Overland Park, Kansas
  - Health East, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Atrial Fibrillation (AF): Patient with a known history of AF who is in AF at the time of study screening.
  1-Lead ECG: All participants will record three single-lead ECGs
  12-Lead ECG: All participants will simultaneously record three 12-lead ECGs
Period: Overall Study
Arm/Group | Atrial Fibrillation (AF) | Normal Sinus Rhythm (SR)
Started | 301 | 301
Completed | 301 | 287
Not Completed | 0 | 14
Not completed — Protocol Violation | 0 | 14

BASELINE CHARACTERISTICS:
Population: 14 participants enrolled as SR but had history of paroxysmal AF and therefore excluded from analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Atrial Fibrillation (AF) | Normal Sinus Rhythm (SR) | Total
Number analyzed (Participants) | 301 | 287 | 588
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.8 (8.62) | 59.5 (17.73) | 66.9 (15.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 159 | 251
  Male | 209 | 128 | 337
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity : Hispanic or Latino | 19 | 57 | 76
  Ethnicity : Not Hispanic or Latino | 282 | 230 | 512
  Race: American Indian or Alaska Native | 2 | 0 | 2
  Race: Asian | 1 | 2 | 3
  Race: Black or African American | 8 | 46 | 54
  Race: Native Hawaiian or Other Pacific Islanders | 0 | 1 | 1
  Race: White | 292 | 236 | 528
  Race: Not Reported | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 301 | 287 | 588

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Software's Rhythm Classification of SR in Agreement to a Physician's Interpretation of a Gold Standard 12-lead ECG
Description: Specificity of rhythm classification
Time Frame: 1 Day
Population: Classifiable Analysis Set: All subjects who had readable/classifiable paired Software and Reference strips were used. This analysis set was used for analyzing the primary endpoints of sensitivity and specificity.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Sinus Rhythm (SR)
Number analyzed (Participants) | 239
Participants | 238
Statistical Analysis 1: Comparison: Normal Sinus Rhythm (SR); H0: Specificity = 92% H1: Specificity > 92 Under the assumption that the true population specificity is 96.5%, 226 subjects who were diagnosed with SR based on the 12-lead ECG reference strip and where the device algorithm classification produced a result of AF or SR was calculated to provide at least 80% power to reject its null hypothesis, using a one-sided type I error of 0.025. To obtain readable waveforms approximately 300 subjects with no known diagnosis of AF were enrolled; Test type: Other; p < 0.0001, 1 sided exact binomial test

2. Primary Outcome: Number of Participants With Software's Rhythm Classification of AF in Agreement to a Physician's Interpretation of a Gold Standard 12-lead ECG
Description: Sensitivity of rhythm classification
Time Frame: 1 Day
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Atrial Fibrillation (AF)
Number analyzed (Participants) | 240
Participants | 236
Statistical Analysis 1: Comparison: Atrial Fibrillation (AF); H0: Sensitivity = 90% H1: Sensitivity > 90% Under the assumption that the true population sensitivity is 95%, 231 subjects who were diagnosed with AF based on the 12-lead ECG reference strip and where the device algorithm classification produced a result of AF or SR was calculated to provide at least 80% power to reject the null hypothesis, using a one-sided type I error of 0.025. To obtain readable waveforms, a minimum of 260 subjects with a known diagnosis of AF were enrolled; Test type: Other; p < 0.0001, 1 sided exact binomial test

3. Secondary Outcome: Number of Participants With Software's Ability to Produce a Clinically Equivalent Waveform in Agreement to a Gold Standard Lead 1 Reference
Description: Number of ECGs that pass a visual overlay
Time Frame: 1 Day
Population: Waveform Assessment Analysis Set: Paired Software and Reference strips collected from subjects were randomly selected. If 6 consecutive paired beats for analysis cannot be found in these strips, they were excluded from further analysis. This analysis set was used for assessing the quality of the clinical waveform.
Measure: Count of Participants; unit: Participants
Arm/Group | Atrial Fibrillation (AF) | Normal Sinus Rhythm (SR)
Number analyzed (Participants) | 61 | 65
Participants | 60 | 65
Statistical Analysis 1: Comparison: Atrial Fibrillation (AF) vs Normal Sinus Rhythm (SR); H0: agreement proportion of visual display= 0.8 H1: agreement proportion of visual display> 0.8 Under the assumption that the true population agreement proportion of visual display was 90%, 88 subjects would provide at least 80% power to reject the null hypothesis using a one-sided type I error of 0.05. To account for obtaining readable waveforms, approximately 140 subjects (70 SR; 70 AF) were randomly selected; Test type: Other; p < 0.0001, 1 sided exact binomial

4. Secondary Outcome: Number of Participants With Software's Ability to Produce a Clinically Equivalent Waveform in Agreement to a Gold Standard Lead 1 Reference
Description: Difference in R-wave amplitudes between the software and gold standard reference
Time Frame: 1 Day
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Atrial Fibrillation (AF) | Normal Sinus Rhythm (SR)
Number analyzed (Participants) | 61 | 65
Participants | 58 | 65
Statistical Analysis 1: Comparison: Atrial Fibrillation (AF) vs Normal Sinus Rhythm (SR); H0: agreement proportion of R wave amplitude = 0.8 H1: agreement proportion of R wave amplitude > 0.8 Under the assumption that the true population agreement proportion of R wave amplitude was 90%, 88 subjects would provide at least 80% power to reject the null hypothesis using a one-sided type I error of 0.05. To account for obtaining readable waveforms, approximately 140 subjects (70 SR; 70 AF) were randomly selected; Test type: Other; p < 0.0001, 1 sided exact binomial

5. Secondary Outcome: Ease of Use
Description: Average ease of use on a 1 (Unable to Use) to 5 (Easiest to Use) scale
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Atrial Fibrillation (AF) | Normal Sinus Rhythm (SR)
Number analyzed (Participants) | 301 | 287
Participants
  1 = Unable to Use | 2 | 1
  2 = Below Average Ease of Use | 4 | 2
  3 = Average Ease of Use | 14 | 16
  4 = Above Average Ease of Use | 41 | 29
  5 = Easiest to Use | 240 | 239

ADVERSE EVENTS:
Time Frame: 1 Day
Description: Adverse Event, Serious Adverse Event or Mortality were assessed/monitored.
Arm/Group | Atrial Fibrillation (AF) | Normal Sinus Rhythm (SR)
All-Cause Mortality (participants affected / at risk) | 0/301 | 0/301
Serious Adverse Events (participants affected / at risk) | 0/301 | 0/301
Other Adverse Events (participants affected / at risk) | 0/301 | 0/301

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT03492554/Prot_SAP_001.pdf